CLINICAL TRIAL: NCT06315530
Title: A Single Center, Randomized Controlled, Open Label Trial Exploring the Regulatory Effect of Telitacicept on Antibody Titers in Primary Antiphospholipid Syndrome Patients Carrying High-risk Antiphospholipid Antibody Profiles
Brief Title: Effect of Telitacicept on Antibody Titers in Primary APS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sh12053
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Antiphospholipid Syndrome (APS)
Keywords: Telitacicept; Antiphospholipid Antibody Profiles
MeSH Terms: conditions — Antiphospholipid Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: SOC+Telitacicept arm (Experimental): Telitacicept 160mg once a week for 48 week as an add-on treatment regimen. SOC treatment includes aspirin and/or vitamin K antagonists (VKA) and/or low molecular weight heparin.
  Interventions: Drug: Telitacicept+SOC; Drug: SOC
- Experimental: SOC arm (Active Comparator): SOC treatment includes aspirin and/or vitamin K antagonists (VKA) and/or low molecular weight heparin.
  Interventions: Drug: SOC

INTERVENTIONS:
Drug: Telitacicept+SOC — 160mg once a week for 48 weeks
  Arms: Experimental: SOC+Telitacicept arm
Drug: SOC — SOC treatment includes aspirin and/or vitamin K antagonists (VKA) and/or low molecular weight heparin.

SUMMARY:
The purpose of this study is to evaluate the regulatory effect of Telitacicept on antibody titers in primary antiphospholipid syndrome patients carrying high-risk antiphospholipid antibody profiles.

DETAILED DESCRIPTION:
This is a single center, randomized controlled trial in Ruijin Hospital. The enrolled patients will be randomized in a 1: 1 ratio to receive either SOC+Telitacicept or SOC treatment.Telitacicept is administered subcutaneously at a dose of 160mg once a week for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Diagnosis of primary APS, meet 2006 Sydney classification criteria or continuously positive for antiphospholipid antibodies within the first 12 months of inclusion (tested at least every 12 weeks), classified as high-risk antiphospholipid antibody spectrum based on the risk of antibody levels, in order to meet at least one of the following conditions: 1. Positive lupus anticoagulant (LAC) (tested according to ISTH guidelines); 2. Two or three types of aPL positivity (lupus anticoagulant, anticardiolipin antibody, and anti-β2 any two or all three types of glycoprotein I antibodies; 3. Or persistent high titer aPL;
* There are no other autoimmune diseases occurring simultaneously;
* According to EULAR recommendations for antiphospholipid syndrome, a stable APS treatment regimen should be adopted;
* Female patients who are not pregnant, breastfeeding, have no fertility potential, or have not undergone contraception.

Exclusion Criteria:

* Patients with a history of malignant tumor in the past 5 years, except for basal cell carcinoma or squamous cell carcinoma of skin or cervical carcinoma in situ treated locally, and there is no evidence of metastasis within 3 years;
* Patients with a history of primary immunodeficiency;
* Serious lack of IgG (IgG level < 400 mg/dL);
* IgA deficiency (IgA level < 10 mg/dL);
* Patients with a current history of infection;
* Patients with a current history of drug or alcohol abuse or dependence, or have a history of drug or alcohol abuse or dependence within 365 days before day 0;
* HIV test is historically positive or HIV screening is positive;
* Hepatitis status;
* Patients with a history of allergic reaction caused by injection of contrast agent, human or mouse protein or monoclonal antibody;
* Patients with other abnormal laboratory values with clinical significance;
* If women with reproductive potential (WCBP) are included, please refer to the following special instructions;
* Patients with concurrent major medical or mental illnesss;
* Patients with diseases of liver, kidney, heart and other important organs,blood and Endocrine system;
* Patients who have been vaccinated with live vaccine in the last month;
* Patients who have participated in any clinical trial within 28 days before the initial screening and/or within 5 times of the half-life of the study compound (whichever is longer);
* Patients who use B-cell targeted therapy drugs within one year, such as rituximab or epratuzumab;
* Patients who use tumor necrosis factor inhibitor and interleukin receptor blocker within one year;
* Patients who use Intravenous gamma globulin (IVIG) and prednisone ≥100mg/d for more than 14 days within one year or plasma exchange;
* Patients with active infection (such as herpes zoster, HIV infection, active tuberculosis, etc.) during the screening period;
* Patients with depression or suicidal thoughts;
* Other conditions that the investigator considers would make the candidate unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with decreased aPL titer at week 48 of treatment | week 48

SECONDARY OUTCOMES:
new thrombotic event | 48 weeks
  any new thrombotic event during Telitacicept treatment
Effects of Telitacicept on the genotype, phenotype, and functional heterogeneity of T and B cells | baseline, week 12, 24, 36, 48
  Application of single-cell RNA sequencing technology (scRNAseq)

OTHER OUTCOMES:
The incidence and severity of adverse events | 48 weeks
  Number and intensity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China